CLINICAL TRIAL: NCT06043843
Title: Effectiveness of a Ramadan-focused Structured Diabetes Tele-education in Reducing Diabetes Complications During Ramadan Fasting in South East Asia
Brief Title: Effectiveness of Focused Tele-education in Reducing Diabetes Complications During Ramadan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Collaborators: Universiti Putra Malaysia (Other); Universiti Teknologi Mara (Other); Universiti Kebangsaan Malaysia Medical Centre (Other); University of Malaya (Other); Universiti Sains Malaysia (Other); Khoo Teck Puat Hospital (Other); Singapore General Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/3137
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus; Fasting; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus; Fasting; Diabetes Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused structured tele-education, medication adjustment and remote monitoring (Active Comparator)
  Interventions: Combination Product: Focused diabetes tele-education and medication adjustment based on guidelines with remote monitoring from trial of fasting from before to throughout Ram
- Control (No Intervention): Standard Care

INTERVENTIONS:
Combination Product: Focused diabetes tele-education and medication adjustment based on guidelines with remote monitoring from trial of fasting from before to throughout Ram — 1. Ramadan-focused online education by physician, specialist nurse, and dietitian via video conferencing
     1. Fasting and exemptions
     2. Self-monitoring of blood glucose
     3. Acute diabetes complications and treatment
     4. Ramadan nutritional plan
     5. Safe physical activity You will be taught to record
     <!-- -->
     1. Meal plans
     2. Physical activities
     3. Blood glucose monitoring, and
     4. Monitoring for diabetes complications Perform a trial fasting day prior to Ramadan.
  2. Medication adjustments will be made according to the Diabetes and Ramadan Alliance guideline as well as individualized modifications based on their HbA1c as follows Baseline HbA1c Recommended dose reduction < 8% 30% 8 to 10% 15% > 10% None
  2) Glucose monitoring
  1. up to 4 times daily Before Ramadan for 1 week During Ramadan After Ramadan for 1 week
  2. uploaded into an online portal for data collection, without remote monitoring.
  Arms: Focused structured tele-education, medication adjustment and remote monitoring

SUMMARY:
Introduction Diabetes is a global emergency with detrimental clinical and financial consequences. Poorly managed diabetes leads to a myriad of serious complications, especially cardiovascular and infectious complications, with consequent increased cost and mortality rate. For Muslims in particular, the annual fasting month of Ramadan is one such period when diabetes control is essential. Adequate adjustments in diabetes management need to be made in line with the allowed mealtimes to avoid the risk of diabetes complications during Ramadan.

Objective Investigators aim to investigate the effectiveness of Ramadan-focused structured diabetes tele-education to reduce diabetes complications during Ramadan fasting for Muslims with diabetes in South East Asia.

Methodology In a parallel group randomized controlled trial, investigators aim to recruit 300 adults with diabetes who are able to fast at least 15 days in Ramadan. You will be randomized to the intervention group comprising of a Ramadan-focused structured diabetes tele-education and control group receiving standard care. You will be reviewed again after Ramadan. The primary outcome is the incidence of hypoglycemia in Ramadan. The secondary outcomes are incidence of other diabetes complications in Ramadan episodes including hyperglycemia, episodes of acute infections, attendances in clinic and emergency department, hospital admissions, and compliance to recommendations for diabetes management during Ramadan.

Clinical Significance The study enables investigators to evaluate Ramadan-focused structured diabetes tele-education to reduce the risk of diabetes complications for a large population during the fasting month.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes planning to fast in Ramadan,

  1. Adults with type 2 diabetes aged at least 21 years old,
  2. Able to fast at least 15 days in Ramadan based on experience of fasting in previous year's Ramadan,
  3. Underlying type 2 diabetes treated with basal insulin and one or more doses of prandial insulin, or at least twice-daily premixed insulin
  4. Performed laboratory tests as per standard care - glycated haemoglobin (HbA1c), serum Low Density Lipoprotein- cholesterol, serum triglycerides, serum High Density Lipoprotein- cholesterol, serum Total cholesterol and serum creatinine
  5. Ability to give informed consent,
  6. Ability to perform self-monitoring blood glucose
  7. Have had diabetes-related clinic visits or hospitalization in the past 10 months.
  8. Have the capacity for video conferencing (internet connection with mobile phone or computer)

Exclusion Criteria:

1. Severe diabetes complications including end-stage renal failure
2. Severe hypoglycemia and hyperglycemic crises within the last 3 months
3. Advanced comorbidities negating the ability to fast
4. Pregnancy
5. Patients on oral medications alone or oral medications plus basal insulin alone
6. Patients on sulfonylureas

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Compare first incidence rate of hypoglycaemia or severe hypoglycemia between intervention and control groups in Ramadan | 4 weeks

SECONDARY OUTCOMES:
Compare the first incidence rate of hypoglycemia or severe hypoglycemia between intervention and control groups in Ramadan when compared to 4 weeks before and 4 weeks post-Ramadan | 12 weeks
Compare the first incidence rate of other complications in Ramadan - hyperglycemia and crises, acute infections, clinic and emergency department attendances and hospital admissions | 12 weeks
Compare the compliance to current Ramadan treatment recommendations for diabetes based on number of blood glucose monitoring during Ramadan | 4 weeks
Compare the compliance to current Ramadan treatment recommendations for diabetes based on number of days of fast terminated in the event of hypoglycaemia or hyperglycemia | 12 weeks
Compare the weight changes after Ramadan as compared to pre-Ramadan weight | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sueziani B Zainudin, Principal Investigator — Sengkang General Hospital
Locations (1):
- Sengkang General Hospital, Singapore, Singapore